CLINICAL TRIAL: NCT02056093
Title: Breathing Pattern Variability, Respiratory Discomfort and Work of Breathing in Proportional Assist Ventilation And Neurally Adjusted Ventilator Assist
Brief Title: Comparison of Proportional Assist Ventilation And Neurally Adjusted Ventilator Assist
Acronym: PAVANAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Matthieu SCHMIDT, Dr, Pierre and Marie Curie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADOREP
Record Dates: First submitted 2013-12-18; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Acute Respiratory Failure
Keywords: NAVA - PAV- Breathing Variability - Asynchrony

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubated patients (Experimental): Intubated patients: The three modes (PSV, PAV, NAVA) will be applied in random order to each mechanically ventilated patient included in the study.
  Interventions: Device: PSV mode; Device: PAV mode; Device: NAVA

INTERVENTIONS:
Device: PSV mode — Application of PSV in all patients
Device: PAV mode — Application of PAV mode in all patients
Device: NAVA

SUMMARY:
In spontaneously breathing mechanically ventilated patients, the adequacy between the patient's demand and the level of respiratory support delivered by the ventilator is a major clinical issue. Neurally adjusted ventilator assist (NAVA) and proportional assist ventilation (PAV) have been developed to adapt the level of assistance to the patient's demand. These two modes have been compared to pressure support ventilation (PSV) but have not been compared to each other.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients.
* Mechanical ventilation for a respiratory reason.
* Expected duration of Mechanical ventilation > 48 hrs.
* Spontaneous breathing.
* Sedations stopped for more than 24 hours.

Exclusion Criteria:

* - Main contra indications to NAVA: gastro-oesophageal surgery in the previous 12 months, oesophageal obstruction, gastro-esophageal bleeding in the previous 30 days, history of esophageal varices, facial trauma or surgery, neuromuscular diseases, individuals with known or suspected phrenic nerve dysfunction.
* Main contra indications to PAV: airway leak, body weight <25 kg, neuromuscular diseases.
* Hemodynamic instability defined as the current administration of vasopressors or inotropic drugs.
* Severe hypoxemia defined as PaO2/FiO2 ratio <200.
* Decision to withhold life-sustaining treatment.
* Pregnant women.
* Minors < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Breathing pattern variability | February 2014
  The coefficient of variation (standard deviation divided by the mean) of the tidal volume (expressed in %)

SECONDARY OUTCOMES:
Patient-ventilator asynchrony | February, 2014
  Prevalence of ineffective efforts and double triggering (expressed as a number of events per minute)

OTHER OUTCOMES:
Electrical diaphragm activity Gas exchange | February 2014
  measured by the NAVA probe

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu SCHMIDT, MD, Principal Investigator — Association pour le Développement et l'Organisation de la Recherche en Pneumologie
Locations (1):
- Service de Pneumologie et de Reanimation médicale, Groupe hospitalier Pitie Salpetriere, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Schmidt M, Kindler F, Cecchini J, Poitou T, Morawiec E, Persichini R, Similowski T, Demoule A. Neurally adjusted ventilatory assist and proportional assist ventilation both improve patient-ventilator interaction. Crit Care. 2015 Feb 25;19(1):56. doi: 10.1186/s13054-015-0763-6. PMID 25879592